CLINICAL TRIAL: NCT03217123
Title: Deep-brain Stimulation in Obsessive-compulsive Disorder
Brief Title: Deep-brain Stimulation in Obsessive-compulsive Disorder: Randomized, Double-blinded Clinical Trial
Acronym: 10/131
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital San Carlos, Madrid (Other)
Responsible Party: Principal Investigator, Juan Antonio Barcia Albacar, Head of Neurosurgery Department, Hospital San Carlos, Madrid
Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: 10/131
Record Dates: First submitted 2017-07-12; First posted 2017-07-13 (Actual); Last update posted 2017-07-18 (Actual); Status verified 2017-07

CONDITIONS: Obsessive-Compulsive Disorder
Keywords: OCD, DBS, fMRI, Y-BOCS, tractography
MeSH Terms: conditions — Obsessive-Compulsive Disorder | interventions — Deep Brain Stimulation

STUDY DESIGN:
Intervention Model Description: The study meets a double-blind, longitudinal design. Stimulation contact was set following a random series known only by the neurosurgeon, with patient, psychiatry and neuropsychology teams blind. Psychiatric assessment was conducted each month, and neuropsychological testing was performed after each activation and washout period
Who Masked: Participant, Care Provider, Investigator
Masking Description: Patients were blind to the study phase (contact and parameters of stimulation).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Deep Brain stimulation (Experimental): After the surgery, a random sequence of contact activations (0 [Nacc],1,2 and 3), including sham (-), was generated for each patient. Each contact was activated using 130 Hz, 60 ms, and 4.5 V for three months (the sham activation was 0 V) following the patient's individual sequence, separated by one month of washout with the generator turned off
  Interventions: Device: Deep Brain stimulation

INTERVENTIONS:
Device: Deep Brain stimulation — Electrical stimulation at subcortical level
  Other Names: Medtronic lead

SUMMARY:
A prospective, randomized, double-blinded study was conducted in 7 OCD patients during which 4 electrode contacts along a striatal axis were stimulated bilaterally. DBS electrode implantation followed a trajectory placing contact zero in nucleus accumbens (a common target for OCD treatment) with more proximal contacts placed in striatal segments defined using projections from prefrontal cortex subdivisions (ventromedial, orbitofrontal, dorsolateral) and anterior cingulate cortex.

DETAILED DESCRIPTION:
Patients Seven patients, three men; aged 21-50 years; average (std) 36.67 (±14.64), and four women; aged 28-46 years; average: 35.25 (±8.14), suffering from treatment-refractory obsessive compulsive disorder participated in this study. All patients scored 30 or higher in the Yale-Brown Obsessive-Compulsive Scale (Y-BOCS). They were considered as candidates to DBS for OCD by two independent psychiatrists. An independent psychiatric surgery committee composed of one neurosurgeon, one psychiatrist and one legal medicine expert agreed surgery indication was appropriate. All patients provided written informed consent. The study had approval from the Hospital Clínico San Carlos ethics committee.

Pre-surgical Neuroimaging Before surgery, all patients underwent 3T Siemens TRIO system (Siemens, Erlangen, Germany) MRI scanning. Patients also performed an OCD symptom provocation task during fMRI scanning using modified version of the MOCSS (Maudsley Obsessive-Compulsive Stimuli Set). During scanning, patients were presented with pictures of 4 classes of provocative stimuli, 50 of each type: 1) contamination/washing, 2) checking, 3) hoarding, 4) symmetry/order. The study comprised 4 'blocks' pertaining to the 4 classes of provocative stimuli. Each block consisted of ten 20-s alternating epochs in which subjects viewed either 10 provocative or 10 neutral pictures (see Supplementary material for a full description). Post-operative computed tomography (CT) scanning was used to determine correct electrode positioning.

Neurosurgical procedure The target was selected for the distal electrode contact (contact zero) to be placed at the NAcc close to the bed nucleus of the stria terminalis: 1.5 mm rostral to the anterior border of the anterior commissure, 4 mm ventral to the AC-PC line and 7 mm lateral to the mid-sagittal plane. Then, the striatum was segmented using the deterministic DTI projections of the three subdivisions of the prefrontal cortex (ventromedial vmPFC, orbitofrontal OFC, dorsolateral DLPFC) plus the anterior cingulate cortex (ACC). A trajectory was planned for placing the rest of the contacts of a Medtronic Model 3391 stimulating macroelectrode at several points along the striatum avoiding the ventricles in such a way that each of the electrode contacts (contacts 1, 2, and 3) was closest to each segment of the striatum corresponding to OFC, DLPFC and ACC.

Deep-Brain Stimulation Protocol After surgery, a random sequence of contact activations (0 [Nacc],1,2 and 3), including sham (-), was generated for each patient. Each contact was activated using 130 Hz, 60 ms, and 4.5 V for three months (the sham activation was 0 V) following the patient's individual sequence, separated by one month of washout with the generator turned off

The study meets a double-blind, longitudinal design. Stimulation contact was set following a random series known only by the neurosurgeon, with patient, psychiatry and neuropsychology teams blind. Psychiatric assessment was conducted each month, and neuropsychological testing was performed after each activation and washout period

Symptom-provocation fMRI analysis Functional imaging data were analyzed using statistical parametric mapping (SPM12; http://www.fil.ion.ucl.ac.uk/spm) employing an epoch-related model. The main symptom(s) for each patient was defined and used to construct a contrast of responses to provocation vs. neutral pictures. The ensuing contrasts were masked with an inclusive prefrontal mask and the statistical parametric map thresholded at P < 0.001 uncorrected. Cluster extent was defined using AlphaSIM (threshold P < 0.05). Note that due to weak responses during symptom activation in patients 4 and 6, the SPMs for these patients were first thresholded at P < 0.01 and 0.005 uncorrected, respectively. After the clinical protocol had ended, the projections to the cortical activated areas on the MOCSS for each patient in their main symptomatic dimension from the striatum were calculated using probabilistic tractography. The connectivity between each of the contacts and the fMRI activations was calculated as the number of fibers of the projection of each contact (sphere of diameter 4 mm around the contact) to the cortical activated areas.

ELIGIBILITY:
Inclusion Criteria:

* Patients suffering from treatment-refractory obsessive compulsive disorder
* Scored 30 or higher in the Yale-Brown Obsessive-Compulsive Scale (Y-BOCS)
* Considered as candidates to DBS for OCD by two independent psychiatrists.
* An independent psychiatric surgery committee composed of one neurosurgeon, one psychiatrist and one legal medicine expert agreed surgery indication was appropriate
* Provide written informed consent.

Exclusion Criteria:

* Any concomitant neurological or psychiatric condition
* Any surgical contraindication

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2011-01-01 (Actual); Primary Completion 2014-12-31 (Actual); Study Completion 2015-06-30 (Actual)

PRIMARY OUTCOMES:
Yale-Brown Obsessive-Compulsive Scale | 2 years
  OCD symptoms scale

SECONDARY OUTCOMES:
Emotion | 2 years
  Depresion and anxiety scores

OTHER OUTCOMES:
Neuropsychology | 2 years
  Neuropsychological scales (A battery of tests, covering the main cognitive domains, was created to assess neuropsychological changes).

CONTACTS AND LOCATIONS:
Overall Officials: Juan A Barcia, MD PhD, Principal Investigator — Hospital San Carlos

IPD SHARING:
Plan to Share IPD: Yes
They will appear in the public report
Supporting Information: CSR
Time Frame: 2017-2018

REFERENCES:
- [Background] Nuttin B, Cosyns P, Demeulemeester H, Gybels J, Meyerson B. Electrical stimulation in anterior limbs of internal capsules in patients with obsessive-compulsive disorder. Lancet. 1999 Oct 30;354(9189):1526. doi: 10.1016/S0140-6736(99)02376-4. PMID 10551504
- [Background] Mataix-Cols D, Wooderson S, Lawrence N, Brammer MJ, Speckens A, Phillips ML. Distinct neural correlates of washing, checking, and hoarding symptom dimensions in obsessive-compulsive disorder. Arch Gen Psychiatry. 2004 Jun;61(6):564-76. doi: 10.1001/archpsyc.61.6.564. PMID 15184236
- [Background] Goodman WK, Foote KD, Greenberg BD, Ricciuti N, Bauer R, Ward H, Shapira NA, Wu SS, Hill CL, Rasmussen SA, Okun MS. Deep brain stimulation for intractable obsessive compulsive disorder: pilot study using a blinded, staggered-onset design. Biol Psychiatry. 2010 Mar 15;67(6):535-42. doi: 10.1016/j.biopsych.2009.11.028. Epub 2010 Feb 8. PMID 20116047
- [Background] Denys D, Mantione M, Figee M, van den Munckhof P, Koerselman F, Westenberg H, Bosch A, Schuurman R. Deep brain stimulation of the nucleus accumbens for treatment-refractory obsessive-compulsive disorder. Arch Gen Psychiatry. 2010 Oct;67(10):1061-8. doi: 10.1001/archgenpsychiatry.2010.122. PMID 20921122